CLINICAL TRIAL: NCT03937518
Title: Strontium Ranelate as New Modality in Treatment of Primary Knee Osteoarthritis
Brief Title: Strontium Ranelate and KOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS 15.09.44
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2018-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — strontium ranelate; Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- strontium ranelate (Other): included 15 patients who received oral strontium ranelate and physiotherapy program. The age of the patients ranged from 50 to 62 years,
  Interventions: Drug: Strontium Ranelate; Other: physiotherapy
- physiotherapy (Other): included 15 patients who received physiotherapy program. The age of the patients ranged from 50 to 62 years
  Interventions: Other: physiotherapy

INTERVENTIONS:
Drug: Strontium Ranelate — Patients received strontium ranelate 2gm (one sachet daily with 50 ml water at bedtime at least 2 h after food), as the compliance of patient assessed by counting number of sachet that patient returns at every visit and safety is assessed by recording adverse effects as blood pressure and heart rate every visit and patients received physiotherapy program in the form of (US therapeutic acoustic radiation and exercise program) 3 times per week for 6 months.
  Ultra sound (US):
  Pulsed ultrasonic waves were delivered at a 1 MHz frequency and at an intensity of 1 watt/ cm2 via a transducer with a diameter of 5 cm and effective radiating area of 3.5 to 5cm² for 9.5 min (
  Arms: strontium ranelate
Other: physiotherapy — Ultra sound (US):
  Pulsed ultrasonic waves were delivered at a 1 MHz frequency and at an intensity of 1 watt/ cm2 via a transducer with a diameter of 5 cm and effective radiating area of 3.5 to 5cm² for 9.5 min (Medserve, England) (Huang et al., 2001). Patients were positioned in a supine position with the affected knee flexed at 90° and the sound head was held stationary over the tibiofemoral joint medial to the patellar tendon to enhance energy penetration into the joint space (White et al., 2007).
  Exercise program:
  The subjects were treated with a group-exercise program composed of a range of motion of all lower limb and 45 min strengthening exercises with 5 min stretching exercises of lower limb muscles 3 times per week under the supervision of the same physiatrist (Fitzgerald and Oatis

SUMMARY:
The present study was carried out on thirty patients with primary knee osteoarthritis. Patients were recruited from Rheumatology and Rehabilitation

Outpatient Clinic at Mansoura University Hospi Patients were divided into two groups:

Group 1: included 15 patients who received oral strontium ranelate and physiotherapy program. The age of the patients ranged from 50 to 62 years, they were 11 females and 4 males. Group 2: included 15 patients who received physiotherapy program. The age of the patients ranged from 50 to 62 years, they were 12 females and 3 males. Written consent was obtained from each participant sharing in the study. This study was approved by the institution research board of faculty of medicine, Mansoura University, code: MS/15.10.08. Inclusion

DETAILED DESCRIPTION:
The present study was carried out on thirty patients with primary knee osteoarthritis. Patients were recruited from Rheumatology and Rehabilitation

Outpatient Clinic at Mansoura University Hospi Patients were divided into two groups:

Group 1: included 15 patients who received oral strontium ranelate and physiotherapy program. The age of the patients ranged from 50 to 62 years, they were 11 females and 4 males. Group 2: included 15 patients who received physiotherapy program. The age of the patients ranged from 50 to 62 years, they were 12 females and 3 males. Written consent was obtained from each participant sharing in the study. This study was approved by the institution research board of faculty of medicine, Mansoura University, code: MS/15.10.08.

InclusionAll patients were subjected to the following:

I. History Taking :

1. Personal History

   * Name, age, sex, residence, marital status.
   * Occupational status.
   * Special habits e.g. smoking status (current/previous).
2. Complaint:

   Taken in the patient's own words with special stress on disease duration.
3. Present history:

   Onset, course and duration of disease. Analysis of complaint Pain: type of pain, site of pain, factors participating/alleviating pain. Swelling. Crepitus. Limitation of movement. Morning and inactivity stiffness, its duration and location. Other joints affected and its pattern of distribution.

   History of other systems affections:

   Neurological symptoms (muscle power and sensation of the lower limbs). Eye symptoms (redness, ulcers and blurred vision). Gastrointestinal tract (GIT) symptoms (diarrhea, heart burn and mucus in the stool). Urinary tract (UT) symptoms (dysuria and frequency). Skin affection (ulcers, erythema, papules and nodules).
4. Past history:

History of surgical operation of knee.

HistoryAssessment of range of motion of the affected knee joint:

For any limitation in the range of motion of the knee joint.

D) Special tests to assess ligaments and menisci:

Varus stress test for lateral collateral ligament. Valgus stress test for medial collateral ligament. Anterior drawer test for anterior cruciate ligament. Posterior drawer test for posterior cruciate ligament.

McMurry's test for menisci.Radiological investigations:

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 40 years with symptoms of knee osteoarthritis

Exclusion Criteria:

rheumatoid arthritis, spondyloarthropathy

Ages: 50 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
change of pain from base line | immediately before intervention,3 monthes after intervention,6 monthes after intervention
  VAS pain is a uni-dimensional tool used to measure pain intensity. It is a 10 cm horizontal line marked every 1 cm. Pain intensity ranges from 0 (no pain, the left end of the line) to 10 (worst possible pain, the right end of the line). The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5- 44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
change of function from base line | immediately before intervention,3 monthes after intervention,6 monthes after intervention
  Patients were assessed before treatment, at 3rd and 6th month after treatment using Western Ontario and McMaster Universities OA index (WOMAC). WOMAC is a self-administered composite questionnaire with three components to assess pain, knee stiffness and difficulty in the activity of daily living. Its first section contains 5 questions about pain, the second section includes 2 questions which assess knee stiffness and the last section is formed of 17 questions that measure the difficulty in the activity of daily living performance.
change of MRI findings from base line | immediately before intervention and 6 monthes after intervention
  Assessment of knee joint by using semi-quantitative MRI by (MOAKS) MRI Osteoarthritis knee score which is performed

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Uninersity Faculty of Medicine, Al Mansurah, Dakahlia Provence, Egypt

IPD SHARING:
Plan to Share IPD: No